CLINICAL TRIAL: NCT00459004
Title: A Dose-Response Relationship Study of SR141716 in Obese Patients
Brief Title: Japanese Dose-Response Study of Rimonabant in Obese Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRI5747
Record Dates: First submitted 2007-04-10; First posted 2007-04-11 (Estimated); Last update posted 2009-04-07 (Estimated); Status verified 2009-04

CONDITIONS: Obesity
Keywords: weight loss
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Rimonabant

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: rimonabant (SR141716)

SUMMARY:
The primary objective is to verify the dose-response relationship of rimonabant on body weight change.

The secondary objectives are to compare the effect of 3 doses of SR141716 to placebo, on body weight loss and on secondary criteria associated with comorbidities, and to evaluate the safety and the pharmacokinetics of SR141716.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index ≥25 kg/m²
* Viceral Fat Area ≥ 100 cm²
* Diet therapy for more than 8 weeks before start of the placebo observation period
* Stable weight (variation < ±3kg within 8 weeks before start of observation period)
* At least 2 criteria of the following 3 comorbidities: Impaired Glucose Tolerance or Type 2 diabetes, Dyslipidemia (hypertriglyceridemia and/or low HDL-choresterol), Hypertension

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 527 (Actual)
Dates: Start 2004-10; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
absolute change in body weight from baseline to Week 24

SECONDARY OUTCOMES:
Efficacy: body weight, visceral fat area, waist circumference, fasting plasma glucose, HbA1c, triglyceride, HDL-cholesterol, blood pressure
Safety:adverse events, laboratory tests, ECGs
Pharmacokinetics: SR141716 plasma trough concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Kohji SHIRAI, Professor, Principal Investigator — Toho University Sakura Medical Center, Japan
Locations (1):
- Sanofi-Aventis, Tokyo, Japan